CLINICAL TRIAL: NCT01642173
Title: Assessment of Coronary Plaque Composition Using Optical Coherence Tomography During Chronic Inhibition of Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activity
Brief Title: Assessment of Coronary Plaque Composition Using Optical Coherence Tomography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Rajiv Gulati, MD Principal Investitgator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-005460
Record Dates: First submitted 2012-06-26; First posted 2012-07-17 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Atherosclerosis; Endothelial Dysfunction; Coronary Small Vessel Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT at baseline (Other): Subjects enrolled in the NIH funded and IRB approved (08-008161) protocol "Lp-PLA2 and Coronary Atherosclerosis in Humans" with a positive diagnosis of coronary artery endothelial dysfunction will be studied using Optical Coherence Tomography during the angiogram at baseline.
  Interventions: Device: Optical Coherence Tomography (C7 XR Dragonfly )
- OCT following 6 month Lp-PLa2 inhibition (Other): Subjects who are enrolled in IRB 10-000044 "Lp-PLA2 and Coronary Atherosclerosis in Humans Aim III" a study in which the investigators are examining the impact of long-term inhibition of Lp-PLA2, with a specific novel inhibitor or placebo, on Lp-PLA2 activity and improvement in coronary endothelial function will be studied using Optical Coherence Tomography during the 6 month return angiogram.
  Interventions: Device: Optical Coherence Tomography (C7 XR Dragonfly )

INTERVENTIONS:
Device: Optical Coherence Tomography (C7 XR Dragonfly ) — Evaluation of the coronary artery using Optical Coherence Tomography utilizing the Dragonfly OCT catheter following a clinically indicated angiogram and endothelial function testing with a positive diagnosis of endothelial dysfunction. The procedure is repeated following 6 months of Lp-PLa2 inhibition or placebo.
  Other Names: C7 XR Dragonfly Optical Coherence Tomography system

SUMMARY:
The investigator's hypothesis is that local activation of the endogenous Lp-PLA2 plays an integral role in early atherosclerosis, and contributes to the mechanism of coronary endothelial dysfunction and to the structural and mechanical properties that characterize plaque vulnerability. Thus, the investigators study will characterize prospectively the correlation between the functional and structural vascular wall properties, and the activity of the Lp-PLA2 pathway.

DETAILED DESCRIPTION:
The present study was a substudy of our National Institute of Health (NIH) funded and Institutional Review Board (IRB) approved (08-008161) protocol "Lp-PLA2 and Coronary Atherosclerosis in Humans" and (10-000044) "Lp-PLA2 and Coronary Atherosclerosis in Humans Aim III" in which the investigators are examining the impact of long-term inhibition of Lp-PLA2, with a specific novel inhibitor, on Lp-PLA2 activity and improvement in coronary endothelial function.

This substudy will use Optical Coherence Tomography (OCT) to quantify alternate features of plaque vulnerability including superficial microcalcification, fibrous cap thickness, and plaque macrophage content at baseline and again at 6 months following Lp-PLA2 inhibition.

The study will provide insight into the role of the endogenous Lp-PLA2 in early coronary atherosclerosis, a potential therapeutic target for early coronary atherosclerosis in humans.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years and < 85 years
* referred to our cardiac catheterization laboratory for coronary vasomotion testing
* are found to have coronary endothelial dysfunction.

Exclusion Criteria:

* these include heart failure
* ejection fraction < 40%
* unstable angina
* myocardial infarction or angioplasty within 6 months prior to entry into the study
* use of investigational agents within 1 month of entry into the study,
* patients who require treatment with positive inotropic agents other than digoxin during the study
* patients with cerebrovascular accident within 6 months prior to entry the study
* significant endocrine, hepatic or renal, disorders
* local or systemic infectious disease within 4 weeks prior to entry into study
* pregnancy or lactation
* mental instability
* Federal Medical Center inmates

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quantification of plaque vulnerability. | change from baseline to six months
  Following recruitment of the total study population and 6-months therapy with the Lp-PLA2 inhibitor or placebo, using Optical Coherence Tomography (OCT) we will quantify alternate features of plaque vulnerability including superficial microcalcification, fibrous cap thickness, and plaque macrophage content comparing baseline and 6 months studies.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Gulati, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States